CLINICAL TRIAL: NCT05611593
Title: A Phase-I, Open Label, Multi-Centre Clinical Study to Assess the Safety, Tolerability and Usability of FOL100 Lotion in Comparison to Oral Finasteride, for the Treatment of Androgenetic Alopecia
Brief Title: Study to Evaluate Safety & Usability of a New Formulation for Male Androgenetic Alopecia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Follicle Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSP-001-FOL1
Record Dates: First submitted 2022-10-19; First posted 2022-11-10 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Androgenic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Finasteride; Tablets

STUDY DESIGN:
Intervention Model Description: Parallel Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOL100 (Experimental): Subjects will apply FOL100 lotion topically in the defined treatment area.
  Interventions: Drug: FOL100
- Propecia 1mg (oral Finasteride) (Active Comparator): Participants will receive1 tablet of Propecia 1mg (oral Finasteride) once daily (q.d)
  Interventions: Drug: Propecia 1Mg Tablet

INTERVENTIONS:
Drug: FOL100 — FOL100 lotion
  Arms: FOL100
Drug: Propecia 1Mg Tablet — Oral Finasteride
  Other Names: Oral Finasteride
  Arms: Propecia 1mg (oral Finasteride)

SUMMARY:
The CSP-001-FOL1 clinical study is aimed to investigate whether local topical administration of FOL100 lotion will be safe for the patient and will not cause local or systemic skin or other adverse events. It is also aimed at indicating effectiveness as compared with oral Finasteride 1mg. In this non-blinded study, each patient will choose his preferred arm (oral finasteride or FOL100 location). During the study, safety and efficacy will be measured as well as usability.

DETAILED DESCRIPTION:
The proposed clinical study aims to test the safety, tolerability and usability of FOL100 compared to the commercially available Finasteride 1mg Propecia in male subjects suffering from AA.

Study endpoints:

Primary Endpoint:

Safety-AE(s) & SAE(s) incidence rate. Secondary Endpoint: Tolerability & usability collecting information on safety, tolerability & usability.

Exploratory Endpoint: Efficacy

1. Mean change in total, vellus and non-vellus hair count, total hair density, cumulative hair diameter and mean hair thickness in the target region.
2. Global photographic assessments.
3. Subject self-assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent will be signed by the subject before starting any study related procedures.
2. Male subject between the ages of 18 to 45 years old.
3. Male subject with mild to moderate vertex male-pattern hair loss, classified as grade III vertex to V, according to the modified Norwood/Hamilton Scale.
4. Subject must be willing to maintain normal shampooing habits and products during the study.
5. Fitzpatrick skin phototype classification of I-IV.
6. Subjects will agree to maintain the same haircut and color throughout the study, with no significant changes that will interfere with study objectives, as determined by the investigator.
7. Ability to understand and cooperate with the investigator and to comply with the requirements of the study protocol.

Exclusion Criteria:

1. Clinically significant abnormal skin findings on the scalp, which in the opinion of the investigator, could interfere with the aim of the study; in particular, abrasion, actinic keratosis, inflammatory disorders, or any other abnormality.
2. Hair transplant surgery or hair weaving.
3. Clinically significant and active physical illness that could interfere with study objectives or may risk patient safety as determined by the Investigator during screening.
4. Ascertained or presumptive hypersensitivity to the active principle and/or any of the formulation ingredients; history of anaphylaxis to drugs or allergic reactions in general, which in the opinion of the investigator may affect subject safety or the outcome of the study.
5. History of local infections of the skin or subcutaneous tissues of the head within 3 months prior to study enrollment.
6. Clinically significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, hematological, endocrine, or neurological diseases, which in the opinion of the investigator may affect subject safety or the outcome of the study.
7. Suspicion of malignancy, including prostate cancer.
8. Subject whose sexual partner(s) is pregnant or plan to become pregnant.
9. Concurrent use of systemic corticosteroids, topical corticosteroids in the area treated in the study, anabolic steroids, or over the counter "hair restorers".
10. Use of any of the following products 1 year for systemic use and 6 months for topical use: minoxidil (topical or oral), zidovudine, cyclosporine, diazoxide, phenytoin, systemic interferon, psoralens, streptomycin, penicillamine ,benoxaprofen, tamoxifen, phenothiazines or cytotoxic agents.
11. Use of oral finasteride or dutasteride, within 18 months prior to enrollment and 6 months prior to enrollment for any topical medication that is considered to affect hair growth.
12. Use of a therapeutic shampoo for hair loss within 1 month prior to enrollment.
13. Light or laser treatment of scalp within 3 months prior to enrollment.
14. Unwilling to undergo a superficial ink marking on the scalp vertex during V0.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Safety of product application | 28 weeks
  Adverse event reporting (local and general)

SECONDARY OUTCOMES:
Tolerability & Usability | 28 weeks
  Subject self-assessment by questionnaire

OTHER OUTCOMES:
Change in hair count | 28 weeks
  Change in total hair count, vellus and non-vellus hair count per cm^2 as assessed by Phototrichogram
Change in total hair density | 28 weeks
  Change in total hair density per cm^2 as assessed by Phototrichogram
Change in hair thickness | 28 weeks
  Change in cumulative diameter and hair thickness per cm^2 as assessed by Phototrichogram
Exploratory Endpoint: Efficacy - self-assess | 28 weeks
  Subject self-assessment by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Solli Brawer, Study Director — Follicle Pharma Ltd
Locations (3):
- Israel (3):
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No